CLINICAL TRIAL: NCT07037953
Title: Association of Serum circ_DLGAP4, lncRNA KCNQ1OT1, and Their Targets miR-9 and SOX7 With Early Diagnosis, Erythropoietin Resistance and Worse Clinical Outcomes of Chronic Kidney Disease: Insights From Hemodialysis Patients
Brief Title: Serum circ_DLGAP4, lncRNA KCNQ1OT1, and Their Targets by Erythropoietin Resistance in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Egyptian Chinese University (Other); Kasr El Aini Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 11551
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis; Chronic Kidney Disease
Keywords: circRNAs; erythropoietin resistance; microRNAs; kidney failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: 60 healthy controls
- non-HD group: 60 CKD patients not receiving hemodialysis (non-HD) group
- HD Group: [60 CKD Grade 5 patients undergoing MHD]

SUMMARY:
Non-coding RNAs have evolved as biomarkers and as phased and specific therapeutic targets for chronic kidney disease (CKD). However, their clinical significance in CKD patients is largely unexplored. Anemia resistant to erythropoietin-stimulating agents (ESAs) is a risk factor for all-cause mortality of CKD patients. This study investigated the potential association of serum circ_DLGAP4, lncRNA KCNQ1OT1, miR-9, and their target SOX7 with the early diagnosis, prognosis, and worse clinical outcomes in CKD patients with different stages, including those on maintenance hemodialysis (MHD). The clinical correlations of these markers in CKD patients were explored; particularly their possible association with ESA resistance in MHD patients.

An analytical observational case-controlled cross-sectional study was conducted on CKD patients. Participants were enrolled to control group [60 healthy controls], on-hemodialysis (non-HD) group [60 CKD Grade 2-4 patients with no hemodialysis], and hemodialysis (HD) Group [60 CKD Grade 5 patients undergoing MHD]. Demographic, clinical, laboratory data, and drug history were recorded. ESA hypo-responsiveness index (EHRI) was calculated. Molecular pathway analysis was conducted using bioinformatics. RT-qPCR and ELISA techniques were used in gene expression and SOX7 protein assays, respectively.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) poses a rising global health challenge, with a median prevalence of 9.5%. In Egypt, an estimated 7.1 million individuals are affected, and the prevalence is expected to increase with the growing incidence of hypertension and diabetes. CKD is now the seventh leading global cause of death, particularly burdening low- and middle-income countries where access to kidney replacement therapy (KRT)-such as dialysis or transplantation-is limited and costly. Early detection and the identification of novel therapeutic targets are essential to delay disease progression and reduce adverse outcomes.

Although urinary albumin-to-creatinine ratio (UACR) and estimated glomerular filtration rate (eGFR) are the clinical standards for CKD diagnosis and staging, both have significant limitations. These include variability, limited sensitivity/specificity, and confounding non-renal factors. Kidney biopsy, while more accurate, is invasive and not routinely feasible. Moreover, controlling traditional risk factors (e.g., hyperglycemia, hypertension) may still fail to prevent progression to end-stage kidney disease (ESKD), which is frequently complicated by anemia and early mortality. This highlights the urgent need for non-invasive, sensitive biomarkers that can aid in diagnosis, prognosis, and treatment guidance.

Non-coding RNAs (ncRNAs), including circular RNAs (circRNAs), long ncRNAs (lncRNAs), and microRNAs (miRNAs), are emerging as promising biomarkers due to their stability in circulation and tissue-specific expression. circRNAs, formed by back-splicing, regulate gene expression by acting as miRNA sponges and are implicated in various kidney disorders, including CKD. Among them, circ_DLGAP4, derived from exons 8-10 of the DLGAP4 gene, has been shown to promote mesangial cell fibrosis and progression of diabetic kidney disease in animal models, though its clinical relevance in human CKD remains unclear.

lncRNAs, such as KCNQ1OT1, also play key roles in CKD pathogenesis by modulating inflammation, fibrosis, and cell proliferation. KCNQ1OT1, located on chromosome 11p15.5, acts as a competing endogenous RNA (ceRNA) for several miRNAs and is associated with renal fibrosis and apoptosis in diabetic nephropathy. Both circ_DLGAP4 and KCNQ1OT1 are known to target miR-9, a miRNA involved in podocyte dysfunction, mitochondrial damage, and cancer-related processes. One of the validated targets of miR-9 is SOX7, a transcription factor involved in vascular development and kidney graft rejection. Despite the theoretical links among these molecules, their integrated roles in CKD pathophysiology are not fully understood.

Hemodialysis (HD) remains a cornerstone for managing advanced CKD. However, patients on maintenance HD (MHD) face high morbidity and mortality. Anemia is nearly universal in ESKD patients and significantly affects their quality of life and survival. Although erythropoiesis-stimulating agents (ESAs) have improved anemia management, a substantial proportion of patients exhibit ESA resistance, leading to increased risks and treatment challenges. ESA hypo-responsiveness-characterized by insufficient hemoglobin response despite high ESA doses-is associated with increased mortality.

Given the biological plausibility and clinical accessibility of ncRNAs in serum, their levels may aid in early detection, prognosis, and treatment stratification in CKD. This study therefore investigated the clinical relevance of serum circ_DLGAP4, KCNQ1OT1, miR-9, and their common downstream target SOX7 across different CKD stages, including patients on MHD. A particular focus was placed on exploring their association with ESA resistance in MHD patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (> 18 years) with a final clinical diagnosis of CKD with a category G2-G5
* mild to severe albuminuria (A1-A3),
* patients with an eGFR < 15 mL/min/1.73 m2 (kidney failure or ESKD) undergoing HD.

Exclusion Criteria:

* Subjects having < 18 years of age,
* non-compliant persons,
* smokers,
* patients with low risk of CKD (category G1),
* kidney transplant recipients,
* individuals in critical conditions, those with acute kidney injury, ischemic heart disease, cancer, or those receiving chemotherapy, or having cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 180 adult participants allocated into 3 groups: control group : 60 healthy volunteers served as controls (age range 33-72 years, 28 males, 32 females), and non-HD group : 60 CKD patients without HD (CKD G2-G4, age range 45-60 years, 29 males, 31 females), and HD group : 60 CKD patients undergoing MHD (CKD G5, age range 44-67 years, 30 males, 30 females).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
SOX7 protein assays | Baseline or Day 1
  Serum SOX7 protein levels determined using Human Transcription Factor SOX7 ELISA kit
circ_DLGAP4 gene expression | Baseline at Day 1
  quantitative PCR, for circ_DLGAP4 according to the kit manufacturer's recommendations.
miR-9-5p gene expression | Baseline at Day 1
  quantitative PCR for miR-9-5p (MIMAT0000441) according to the manufacturer's kit recommendations.

SECONDARY OUTCOMES:
ESA hypo-responsiveness index (EHRI) | Baseline or at Day 1
  calculated using the equation ERI = [dose of ESA (IU/ week)]/[Hb (g/dL) × body weight (kg)]

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sabry, PhD, Principal Investigator — Clinical pharmacy department, Faculty of pharmacy and drug technology, Egyptian Chinese University
Locations (1):
- Unit of Renal Failure Therapy and Surgery, Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo, Egypt, and the Hemodialysis Unit, New Cairo Specialized Hospital, Cairo, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
will be available upon reasonable request